CLINICAL TRIAL: NCT01908309
Title: Contrast-inDuced nephRotoxicity as Assessed by the Cystatin-modified KIdney Load-to-DAmage RElationship
Brief Title: Contrast-inDuced nephRotoxicity as Assessed by the KIdney Load-to-DAmage RElationship
Acronym: DrKILDARE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Azienda Sanitaria Locale 9, Grosseto (Other Government)
Responsible Party: Principal Investigator, Ugo Limbruno, MD, PhD, Azienda Sanitaria Locale 9, Grosseto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K-3
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Contrast Induced Acute Kidney Injury
Keywords: acute kidney injury; contrast media; cystatin-C
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iodixanol (Active Comparator): Patients randomized to coronary angiography/angioplasty with Iodixanol 320
  Interventions: Drug: Iodixanol 320
- Iobitridol (Active Comparator): Patients randomized to coronary angiography/angioplasty with Iobitridol 350
  Interventions: Drug: Iobitridol 350

INTERVENTIONS:
Drug: Iobitridol 350
  Arms: Iobitridol
Drug: Iodixanol 320
  Arms: Iodixanol

SUMMARY:
We previously demonstrated that the slope of the relationship plotting individual iodine loads against contrast-induced serum creatinine changes ( the load-to-damage relationship, LDR) characterizes the intrinsic nephrotoxicity of the contrast. Aim of the present study is to compare, through the assessment of the LDR slope, the intrinsic nephrotoxicity of two different contrast media using serum cystatin-C changes as the LDR dependent variable.

DETAILED DESCRIPTION:
We previously demonstrated that the slope of the relationship plotting individual iodine loads against contrast-induced serum creatinine changes ( the load-to-damage relationship, LDR) characterizes the intrinsic nephrotoxicity of the contrast and it may allow for reliable comparative evaluations among small sized study groups randomized to different contrast media. The aim of the present study is to compare, through the assessment of the LDR slope, the intrinsic nephrotoxicity of two different contrast media using serum cystatin-C changes as the LDR dependent variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidate to coronary angiography and/or angioplasty and
* Baseline creatinine clearance < 60 ml/min

Exclusion Criteria:

* Patients with STEMI
* Patients with shock
* Known allergy to contrast media
* Prior contrast administration within 1 month
* Current use of nonsteroidal anti-inflammatory drugs

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Slope of LDR (as assessed by serum cystatin-C changes) | 48 hours
  Slope of the relationship plotting individual iodine loads against serum cystatin-C changes at 48 hours after catheterization

SECONDARY OUTCOMES:
Slope of LDR (as assessed by serum creatinine changes) | 72 hours
  Slope of the relationship plotting individual iodine loads against serum creatinine changes at 72 hours after catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Misericordia Hospital, ASL 9, Grosseto, Italy

REFERENCES:
- [Background] Limbruno U, Picchi A, Micheli A, Calabria P, Cortese B, Brizi G, Severi S, De Caterina R. Refining the assessment of contrast-induced acute kidney injury: the load-to-damage relationship. J Cardiovasc Med (Hagerstown). 2014 Jul;15(7):587-94. doi: 10.2459/JCM.0b013e3283638e56. PMID 23811842